CLINICAL TRIAL: NCT02195167
Title: A Safety, Tolerability, Pharmacokinetic, and Pharmacodynamic Evaluation of Single Oral Doses of SEP-225289 in Subjects 6 to 17 Years of Age With Attention Deficit Hyperactivity Disorder
Brief Title: Dasotraline SEP360-105 Pediatric PK/PD Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SEP360-105
Record Dates: First submitted 2014-07-17; First posted 2014-07-21 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: Pediatric Attention Deficit Hyperactivity Disorder
MeSH Terms: interventions — 4-(3,4-dichlorophenyl)-1,2,3,4-tetrahydronaphthalen-1-amine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dasotraline (Experimental): Dasotraline 1 mg, 2 mg, 4 mg, 8 mg, 12 mg, 16 mg, 20 mg, 24 mg, 28 mg, 32 mg once daily. The planned dose for the first cohort is 1mg. There will be no more than a 2-fold increase in dose increase in dose between consecutive dose cohorts up to 8 mg, and dose cohorts beyond the 8 mg level will increment no more than 4mg. The maximum dose will not exceed 32mg." The language should precede the text that is currently there
  Interventions: Drug: Dasotraline 1 mg, 2 mg, 4 mg, 8 mg, 12 mg, 16 mg, 20 mg, 24 mg, 28 mg, 32 mg once daily

INTERVENTIONS:
Drug: Dasotraline 1 mg, 2 mg, 4 mg, 8 mg, 12 mg, 16 mg, 20 mg, 24 mg, 28 mg, 32 mg once daily — Dasotraline 1 mg, 2 mg, 4 mg, 8 mg, 12 mg, 16 mg, 20 mg, 24 mg, 28 mg, 32 mg once daily. The planned dose for the first cohort is 1mg. There will be no more than a 2-fold increase in dose increase in dose between consecutive dose cohorts up to 8 mg, and dose cohorts beyond the 8 mg level will increment no more than 4mg. The maximum dose will not exceed 32mg." The language should precede the text that is currently there

SUMMARY:
Pediatric PK study of SEP-225289 (Dasotraline)

DETAILED DESCRIPTION:
To characterize the pharmacokinetics (PK) and assess safety and tolerability of a range of single oral doses of SEP-225289 in subjects 6 to 17 years old with ADHD

ELIGIBILITY:
Inclusion Criteria:

Subject, male or female, must be between 6 and 17 years of age, inclusive, at the time of consent. Note: Subjects who are 17 years of age at time of consent must not have a birthday within the following 4 weeks in order to be eligible for the study.

* Subject meets Diagnostic and Statistical Manual of Mental Disorders Fourth Edition; Text Revision (DSM-IV-TR) criteria for a primary diagnosis of ADHD (inattentive, hyperactive, or combined subtype) established by a comprehensive psychiatric evaluation that reviews DSM-IV-TR criteria prior to Screening. Diagnosis is confirmed at Screening using Mini International Neuropsychiatric Interview for Children and Adolescents (MINI-KID).
* Subject's parents/legal guardians must give written informed consent, including privacy authorization, prior to study participation. The subject will complete an informed assent prior to study participation. Note: Informed consent will be obtained from both parents unless one parent is deceased, unknown, incompetent, or when one parent has legal responsibility for the care and custody of the child.
* Subject and the subject's parents/legal guardians must be judged by the investigator to be willing and able to comply with the study procedures and visit schedules, including venipuncture, overnight stay (recommended for parent/legal guardian to remain overnight with the subject), and follow-up visits.
* Subject, if female, must not be pregnant or breastfeeding, and if ≥ 8 years of age must have a negative serum pregnancy test at screening.
* Female subjects of childbearing potential and male subjects with female partners of childbearing potential must agree to use an effective and medically acceptable form of birth control throughout the study period.
* Subject must be in general good health (defined as the absence of any clinically relevant abnormalities as determined by the investigator) based on screening physical and neurological examinations, medical history, and clinical laboratory values (hematology, chemistry, and urinalysis). Note: If any of the hematology, chemistry, or urinalysis results are not within the laboratory's reference range, then the subject can be included only if the investigator determines the deviations to be not clinically relevant.
* Subject is within 3rd to 97th percentile for gender specific body mass index (BMI)-for-age from the World Health Organization (WHO) growth charts (Appendix VI) and weighs at least 25 kg.
* Subject must report a history of being able to swallow capsules.
* Subject and subject's parents/legal guardians must be able to fully comprehend the informed consent/assent form, understand all study procedures, and be able to communicate satisfactorily with the investigator and study coordinator.

Exclusion Criteria:

Subject or parents/legal guardians have daily commitments during the study that would interfere with attending study visits.

* Subject has any clinically significant unstable medical abnormality, chronic disease, or a history of a clinically significant abnormality of the cardiovascular,gastrointestinal, respiratory, hepatic, or renal systems, or a disorder or history of a condition (eg, malabsorption, gastrointestinal surgery) that may interfere with drug absorption, distribution, metabolism, or excretion.
* Subject has a history or presence of abnormal ECGs, which in the investigator's opinion is clinically significant. Screening ECGs will be centrally over-read, and eligibility will be determined based on the over-read report.
* Subject has a documented history of Bipolar I or II Disorder, major depression, conduct disorder, oppositional defiant disorder, generalized anxiety disorder (other than obsessive-compulsive disorder) or any history of psychosis, that has been the primary focus of treatment at any time during the 12 months prior to screening.
* Subject has organic brain disease, for example, traumatic brain injury residua, or a history of febrile seizures. Subjects taking anticonvulsants for seizure control currently or within the past 2 years are not eligible for study participation.
* Subject answers "yes" to "Suicidal Ideation" item 4 (active suicidal ideation with some intent to act, without specific plan) or item 5 (active suicidal ideation with specific plan and intent) on the C-SSRS Children's Lifetime/Recent assessment at screening. Subjects who have significant findings for suicidal ideation upon completion of the C-SSRS must be referred to the investigator for follow-up evaluation.
* Subject has any history of attempted suicide.
* Subject does not tolerate venipuncture or has poor venous access that would cause difficulty for collecting blood samples.
* Subject has a history of severe allergies to more than 1 class of medications or multiple adverse drug reactions.
* Subject has history of exposure to stimulants with intolerable side effects.
* Subject has taken any antipsychotic medication within 8 weeks of Visit 1 (Screening).
* Subject is taking any psychotropic medication, including health-food supplements with purported central nervous system activity (eg, St. John's Wort, melatonin), must have a washout equal to a minimum of 5 half lives of that medication prior to Visit 2. If the half life of a medication is unknown, for example, herbal products, then the subject should have a 28 day medication washout.
* Subject is currently taking an antidepressant medication (eg, bupropion, selective serotonin reuptake inhibitor [SSRI]/ serotonin norepinephrine reuptake inhibitor [SNRI], monoamine oxidase [MAO] blocker, tricyclic, etc).
* Subject or subject's family anticipates a move outside the geographic range of the investigative site during the study period, or plans extended travel inconsistent with the recommended visit interval during study duration.
* Subject has a history of, or current malignancy except for non melanoma skin cancer.
* Subject has a positive screening test for Hepatitis B surface antigen, Hepatitis C antibody, or human immunodeficiency virus (HIV)-1 or HIV-2.
* Subject has participated in any investigational study within 30 days prior to screening or is currently participating in another clinical trial.
* Subject has a history of substance abuse or drug dependence (excluding nicotine and caffeine) within the 12 months prior to screening, as defined by the DSM IV TR criteria or has a positive urine drug screen (UDS), cotinine test, or breath alcohol test at Visit 1.
* Subject is taking any disallowed medications for chronic treatment.
* Subject has experienced significant blood loss within 60 days or has donated plasma within 72 hours prior to Visit 1 or intends to donate blood or undergo elective surgery within 30 days following Visit 2.
* Subject has a history of allergic reaction or has a known or suspected sensitivity to any substance that is contained in the study drug formulation.
* Subject is a relative of an investigational site staff member.
* Subject is, in the opinion of the investigator, unsuitable in any other way to participate in this study.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 105 (Actual)
Dates: Start 2014-07; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Maximum concentration (Cmax), tmax, t1/2, area under the concentration from time zero to infinite time (AUC0-inf), and AUC0-last. | 0-51 Days
Incidence of AEs, SAEs, and discontinuation due to AE | 0-51 Days
Clinical Global Impressions-Severity of Illness (CGI-S) score and Columbia Suicide Severity Rating Scale (C-SSRS) evaluation. | 0-51 Days
Absolute values-changes from baseline in clinical laboratory tests, vital signs, orthostatic changes, and 12-lead electrocardiograms (ECGs). | 0-51 Days

SECONDARY OUTCOMES:
Apparent clearance (CL/F), apparent volume of distribution (Vz/F), and terminal elimination rate constant (λz). | 0-51 Days
Time to maximal reduction of plasma DHPG, percent maximal reduction of plasma DHPG concentration relative to baseline, minimal observed plasma DHPG concentration postdose, and time to minimal observed plasma DHPG concentration postdose. | 0-51 Days

CONTACTS AND LOCATIONS:
Overall Officials: Dasotraline Medical Director, MD, Study Director — Sumitomo Pharma America, Inc.
Locations (12):
- United States (12):
  - Woodland International Research Group, Little Rock, Arkansas
  - MCB Clinical Research Centers, LLC, Colorado Springs, Colorado
  - Palm Springs Research Institute, Hialeah, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - iResearch Atlanta, LLC, Decatur, Georgia
  - Louisiana Research Associates, Inc, New Orleans, Louisiana
  - Wake Research, Raleigh, North Carolina
  - IPS Research Company, Oklahoma City, Oklahoma
  - Cutting Edge Research Group, Oklahoma City, Oklahoma
  - Clinical Trials of Texas, Inc. (CTT), San Antonio, Texas
  - Road Runner Research, San Antonio, Texas
  - Aspen Clinical Research, Orem, Utah